CLINICAL TRIAL: NCT04302662
Title: A Multicenter, Open-label Phase 2 Study With Escalating Doses of MS1819-SD on Top of a Stable Dose of PPEs, to Investigate the Efficacy and Safety of This Combination for the Compensation of Severe Exocrine Pancreatic Insufficiency in CF Patients Not Fully Compensated With Only PPEs
Brief Title: Phase 2 Combination Study With Escalating Doses of MS1819-SD on Top of a Stable Dose of PPEs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AzurRx SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS1819/18/02
Record Dates: First submitted 2020-03-04; First posted 2020-03-10 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis Gastrointestinal Disease; Cystic Fibrosis of Pancreas
Keywords: Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Intervention Model Description: Sequential assignment: eligible patients will be receiving increased doses from lower, middle to upper range of MS1819-SD on top of a stable dose of PPEs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: MS1819-SD — Patients will receive increasing doses from the lowest to a maximum dose of MS1819-SD on top of a stable dose of PPEs. The total treatment phase will range from 39 to 51 days.

SUMMARY:
This is a Phase 2 study sponsored by AzurRx SAS and involves testing of a new medication for the compensation of exocrine pancreatic insufficiency (EPI) caused by cystic fibrosis (CF). The new medication is called MS1819 spray dried (MS1819-SD) which is a lipase produced by the Lip2 gene of Yarrowia lipolytica using recombinant DNA technology.

The primary purpose of this study is to investigate the efficacy and safety of escalating doses of study drug on top of a stable dose of PPEs in CF patients who are not fully compensated by PPEs only.

This enzyme has demonstrated an appropriate profile to compensate the pancreatic lipase (enzyme) deficiency that is common in CP (chronic pancreatitis) and CF patients.

The design of the study is open-label, meaning that all eligible patients will receive the study drug MS1819-SD. The study drug dose will increase throughout the study during dose escalation visits in each treatment period; study includes a total of three treatment periods.

The total duration of the MS1819-SD treatment phase is of 39-51 days. The total duration of patient participation in the study is of 69-81 days. Approximately 24 patients will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form.
2. Age > 12 years at the time of screening
3. Male or female.
4. Under stable dose of PPE ≥ 1 month. Stable dose is defined as dose of medication not changed during this time period and the medication must be commercially available and be administered in the recommended dose range.
5. A nutritional status as defined by:

   1. BMI ≤ 22.0 kg/m2 for female patients
   2. BMI ≤ 23.0 kg/m2 for male patients
   3. BMI ≤ 50th percentile for patients 12 to < 18 years of age.
6. Cystic fibrosis, based on 2 clinical features consistent with CF in the opinion of the investigator AND sweat chloride concentration > 60 mmol/L by pilocarpine iontophoresis.
7. Faecal pancreatic elastase-1 < 100 µg/g of stools at screening.
8. Baseline CFA < 80% with a maximum daily dose of 10,000 lipase units/kg/day.
9. Clinically stable with no documented evidence of significant respiratory symptoms that would require administration of intravenous antibiotics, oxygen supplementation, or hospitalization within the 30 days of screening.
10. Male and female patients, if of childbearing potential, must use a reliable method of contraception during the study. A reliable method of birth control is defined as one of the following: oral or injectable contraceptives, intrauterine device, contraceptive implants, tubal ligation, hysterectomy, or a double-barrier method (diaphragm with spermicidal foam or jelly, or a condom), abstinence or vasectomy. Periodic abstinence (calendar, symptothermal, or post-ovulation methods) is not an acceptable method of contraception. The preferred and usual lifestyle of the patient must also be evaluated in determining if sexual abstinence is a reliable method of birth control.
11. Be considered as reliable and capable of adhering to the protocol, according to the judgment of the investigator.

Exclusion Criteria:

1. Established or suspected fibrosing colonopathy.
2. Total or partial gastrectomy.
3. A history of solid organ transplant or significant surgical resection of the bowel; significant resection of the bowel is defined as any resection of the terminal ileum or ileocecal valve. Patients who have had qualitative, long-term changes in nutritional status after any other bowel resection (eg, increased of new need for pancreatic enzyme supplementation compared with preoperative status to maintain the same nutritional status) should also be excluded.
4. Any chronic diarrheal illness unrelated to pancreatic insufficiency (eg, infectious gastroenteritis, sprue, inflammatory bowel disease)
5. Known hypersensitivity or other severe reaction to any ingredient of the investigational medicinal product (IMP).
6. Bilirubin > 1.5 times upper limit normal (ULN).
7. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times ULN.
8. Alkaline phosphatase (ALP) > 5 times ULN.
9. Gamma glutamyltransferase (GGT) > 5 times ULN.
10. Signs and/or symtoms of liver cirrhosis or portal hypertension (eg, splenomegaly, ascites, esophageal varices), or documented liver disease unrelated to CF
11. Patients with a known allergy to the stool marker.
12. Feeding via an enteral tube during 6 months before screening
13. Routine use of anti-diarrheals, anti-spasmodics, or cathartic laxatives, or a change in chronic osmotic laxatives (eg, polyethylene glycol) regimen in the previous laxative therapy within the last 12 months before screening
14. History of severe constipation with < 1 evacuation/week under appropriate laxative therapy within the last 12 months before screening.
15. Documentation of distal intestinal pseudo-obstruction syndrome within the last 12 months before screening.
16. Forced Expiratory Volume ≤ 30% at the screening visit.
17. Lactation or known pregnancy or positive pregnancy test at both screening and baseline for women of childbearing potential.
18. Participation in another clinical study involving an IMP within 30 days before inclusion or concomitantly with this study.
19. Poorly controlled diabetes according the investigator's judgement.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Coefficient of fat absorption | 15 days
  determination of fat absorption based on fat intake and fat excretion over 3 days on high fat meal
Adverse Events | 81 days
  AE, SAE, SUSAR, immunoallergic reactions

SECONDARY OUTCOMES:
Weight of stools | 15 days
  evaluation of changes in weight of stools from baseline (PPEs only) to each treatment period
number of daily evacuations | 15 days
  evaluation of changes in daily evacuations from baseline (PPEs only) to each treatment period
Steatorrhea, | 15 days
  evaluation of changes in steatorrhea from baseline (PPEs only) to each treatment period
Creatorrhea | 15 days
  evaluation of changes in creatorrhea from baseline (PPEs only) to each treatment period
Body weight | 15 days
  evaluation of changes in body weight from baseline (PPEs) to each treatment period
Consistency of stools | 15 days
  evaluation of consistency of stools from baseline (PPEs) to each treatment period

CONTACTS AND LOCATIONS:
Locations (10):
- Hungary (4):
  - Országos Korányi TBC és Pulmonológiai Intézet Cisztás Fibrózis Részleg, Budapest
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktatókórház, Gyermekegészségügyi Központ, Miskolc
  - Somogy Megyei Kaposi Mór Oktató Kórház, Mosdósi telephelye Mosdósi Gyermekrehabilitációs és Gyermekpulmonológiai Egység, Mosdós
  - Tüdőgyógyintézet Törökbálint Gyermekpulmonológiai Osztály és Szakrendelés, Törökbálint
- Turkey (Türkiye) (6):
  - Çukurova University School of Medicine, Adana
  - Hacettepe University School of Medicine, Ankara
  - Akdeniz University School of Medicine, Antalya
  - Cerrahpasa University School of Medicine, Istanbul
  - Mamara University School of Medicine, Istanbul
  - Necmettin Erbakan University,Meram School of Medicine, Konya

IPD SHARING:
Plan to Share IPD: Undecided